CLINICAL TRIAL: NCT03421847
Title: Study of Rotatory Vestibular Tests in Major Depression Patients and Healthy Control Subjects.
Status: Completed | Type: Observational
Sponsor: Vest Brain,Centro de Estudios Neurovestibulares (Other)
Collaborators: Centro de Medicina Aeroespacial. (Unknown)
Responsible Party: Sponsor
Other Study IDs: ROTDEPR01
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Depression; Vestibular Disorder
Keywords: depression; vestibular disorder; rotatory test; electronystagmography
MeSH Terms: conditions — Depression; Vestibular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Major Depression Group: We will measure the vestibular activity of Major depression patients with Rotatory Test and electronystagmography
  Interventions: Diagnostic Test: Rotatory vestibular test
- Healthy Control Group: We will measure the vestibular activity of Healthy subjects with Rotatory Test and electronystagmography.
  Interventions: Diagnostic Test: Rotatory vestibular test

INTERVENTIONS:
Diagnostic Test: Rotatory vestibular test — We will measure Depression and Healthy subjects vestibular activity by Rotatory Vestibular tests

SUMMARY:
This study evaluates the vestibular activity in major depression patients and healthy controls using the rotatory test and electronystagmography.

DETAILED DESCRIPTION:
Previous studies showed abnormal vestibular activity in major depression patients using caloric vestibular tests. The present study investigates the vestibular response to vestibular rotatory tests in major depression subjects and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* male and females adults (18 years or older)
* met the Diagnosing and Statistical Manual of Mental Disorders (DSM-IV-R, American Psychiatric Association, 2000) criterion.
* had a score of 12 or more in the Hamilton Rating Scale, 21 items for Depression.
* with or without actual pharmacological treatment, except benzodiazepines that were suspended 24 hours before the rotary test when corresponding.

Exclusion Criteria:

* pregnant women
* neurologic disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Depression Group patients were selected by psychiatrists from the ambulatory Mental Health consult of the Hospital; the Control Group included 20 healthy volunteers, composed by desk workers from the center.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2005-07-01 (Actual); Primary Completion 2006-12-15 (Actual); Study Completion 2006-12-15 (Actual)

PRIMARY OUTCOMES:
Vestibular Activity | Vestibular rotatory test for each participant is about 50- 60 minutes. One rotatory test per participant.
  The primary outcome corresponds to the vestibular activity. The vestibular stimulation provided by the rotatory chair is sensed by the inner ear´s vestibular receptors and generates reflex ocular movements(Vestibulo Ocular Reflex) registrated by electronystagmography. The main outcome corresponds to the asymmetry of the vestibular activity between both ears.

IPD SHARING:
Plan to Share IPD: Yes
We plan to share all collected vestibular data of IPD after 6 months of publication.
Supporting Information: Analytic Code
Time Frame: Data will be available after 6 months of publication undefined.